CLINICAL TRIAL: NCT01289327
Title: Propofol Versus Midazolam Plus Alfentanil for Sedation During Flexible Bronchoscopy: Respiratory Depression Comparison Inspected by Cutaneous Carbon Dioxide Tension Level
Brief Title: Propofol Versus Midazolam+Alfentanil for Sedation During Bronchoscopy: Comparison by Cutaneous Carbon Dioxide Tension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Mordechai R Kramer, MD,Professor, Rabin Medical Center/Clalit
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5634
Record Dates: First submitted 2011-01-16; First posted 2011-02-03 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2010-12

CONDITIONS: Lung Disease
MeSH Terms: conditions — Lung Diseases | interventions — Propofol; Midazolam; Alfentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propofol (Active Comparator)
  Interventions: Drug: Sedation with Propofol or Midazolam+Alfentanil for FFB
- midazolam+alfentanil (Active Comparator)
  Interventions: Drug: Sedation with Propofol or Midazolam+Alfentanil for FFB

INTERVENTIONS:
Drug: Sedation with Propofol or Midazolam+Alfentanil for FFB — Sedation was started with intravenous injection of a bolus of 2-4 mg midazolam and 0.5 mg alfentanil or 20-50 mg propofol. It was maintained with intermittent boluses of 1-3 mg intravenous midazolam or 0.5 mg intravenous alfentanil, according to clinical judgment, or with boluses of 10-20 mg intravenous propofol, administered at short intervals (~2 minutes) or according to clinical judgment.
  Other Names: diprivan; midazolam; alfentanil

SUMMARY:
Although propofol is a popular agent for sedation during flexible bronchoscopy, some clinicians have raised concerns that it may cause greater respiratory drive reduction than more common drugs. However, this factor is difficult to accurately examine with pulse oximetry. The introduction of a novel device that noninvasively measures carbon dioxide (CO2) levels can help to resolve this controversy. The aim of this study is to evaluate the safety of conscious sedation with midazolam+alfentanil compared to propofol.

DETAILED DESCRIPTION:
Methods: The study group included 115 patients undergoing flexible fiberoptic bronchoscopy(FFB). Patients were randomly assigned by a computer before the procedure to receive sedation with midazolam+alfentanil or propofol. Local anesthesia was induced by application of 2% lidocaine to the oropharynx. Sedation was started with intravenous injection of a bolus of 2-4 mg midazolam and 0.5 mg alfentanil or 20-50 mg propofol. It was maintained with intermittent boluses of 1-3 mg intravenous midazolam or 0.5 mg intravenous alfentanil, according to clinical judgment, or with boluses of 10-20 mg intravenous propofol, administered at short intervals (~2 minutes) or according to clinical judgment.

In all cases, monitoring included continuous electrocardiography, pulse oximetry, and automated noninvasive blood pressure recordings every 5 minutes. In addition, percutaneous carbon dioxide tension (PcCO2) was measured with a cutaneous digital sensor (Sentec AG, Therwil, Switzerland) that was placed on the earlobe prior to the procedure. It was removed when the patient left the bronchoscopy suite.

During the procedure, all patients received supplemental nasal oxygen at 2-5 L min-1. Significant hypoxemia, defined as functional oxygen saturation (SpO2) of 90%, was treated initially with jaw support. If it lasted more than few seconds, a naso/oropharyngeal tube was inserted or supplemental oxygen was delivered via face mask at 10 L min-1. The duration of bronchoscopy was calculated from the administration of sedation until the flexible bronchoscope was removed from the tracheobronchial tree.

Percutaneous carbon dioxide tension, blood oxygenation, heart rate, and blood pressure were compared between the groups.

A questionnaire evaluating pain and discomfort by Visual Analog Scale was completed by the patient when awake after the procedure.(~30 minutes after the end of the procedure

ELIGIBILITY:
Inclusion Criteria:

* The study group consisted of patients scheduled for flexible bronchoscopy under local anesthesia with sedation at a tertiary medical center.

Exclusion Criteria:

* Inability or refusal to provide informed consent, age less than 18 years, bronchoscopy through an artificial airway, and allergy to soya or to one of the sedative drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Percutaneous carbon dioxide tension | From the beginning of fiberoptic bronchoscopy until 10 minutes after the end of the procedure (average time of fiberoptic bronchoscopy ~ 15 minutes)
  Continues measurements (record every 4 second)
oxygen saturation | From the beginning of fiberoptic bronchoscopy until 10 minutes after the end of the procedure (average time of fiberoptic bronchoscopy ~ 15 minutes)
  Continues measurements (record every 4 second)
heart rate | From the beginning of fiberoptic bronchoscopy until 10 minutes after the end of the procedure (average time of fiberoptic bronchoscopy ~ 15 minutes)
  Continues measurements (record every 4 second)
non invasive blood pressure | From the beginning of fiberoptic bronchoscopy until 10 minutes after the end of the procedure (average time of fiberoptic bronchoscopy ~ 15 minutes)
  every 5 minutes

SECONDARY OUTCOMES:
A questionnaire evaluating pain and discomfort | ~30 minutes after the end of the procedure
  A questionnaire evaluating pain and discomfort by Visual Analog Scale was completed by the patient when awake after the procedure.(~30 minutes after the end of the procedure)
Oxygen supplementation | From the beginning of fiberoptic bronchoscopy until 10 minutes after the end of the procedure (average time of fiberoptic bronchoscopy ~ 15 minutes)
  Significant hypoxemia, defined as functional SpO2 of 90%, was treated initially with jaw support. If it lasted more than few seconds, a naso/oropharyngeal tube was inserted or supplemental oxygen was delivered via face mask at 10 L min-1.
  The percentage of patients who needed supplemental oxygen was evaluated
Naso/oropharyngeal tube insertion | From the beginning of fiberoptic bronchoscopy until 10 minutes after the end of the procedure (average time of fiberoptic bronchoscopy ~ 15 minutes)
  Significant hypoxemia, defined as functional SpO2 of 90%, was treated initially with jaw support. If it lasted more than few seconds, a naso/oropharyngeal tube was inserted or supplemental oxygen was delivered via face mask at 10 L min-1
  The percentage of patients who needed Naso/oropharyngeal tube insertion was evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai R Kramer, MD,Professor, Principal Investigator — Head, Pulmonary Institute , Rabin Medical center, Beilinson Hospital, Petach Tikva, 49100 Israel
Locations (1):
- Rabin Medical center, Beilinson Hospital, Petah Tikva, Israel